CLINICAL TRIAL: NCT06102876
Title: Feasibility of Physical Activity in Older Adults With Haematological Malignancies: ACCES Study (Aging & CanCer : Exercise as a Solution)
Brief Title: Feasibility of Physical Activity in Older Adults With Haematological Malignancies: ACCES Study
Acronym: ACCES
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0409
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Geriatric; Haematologic Neoplasm
Keywords: older adults; cancer; physical activity; deconditioning; sedentarity; aging-well
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Physical activity (PA) program — The PA program is specific for each patient according to their mobility profile assessed using a decision tree comprising 3 tests: 1) the number of repetitions in the 30-second sit-to-stand test, 2) the score in the Short Physical Performance Battery (SPPB) test and 3) grip strength. The PA program has to be performed once daily.

SUMMARY:
The aim of this study is to implement a simple and unsupervised home-based physical activity (PA) program for cancer patients in 2 oncogeriatric units in Toulouse Hospital (day hospital and week hospital).

DETAILED DESCRIPTION:
Cancer treatments can cause side effects such as fatigue and reduced muscle function. Studies have shown the benefits of physical activity, including reduced fatigue and improved quality of life. Moreover, PA is often recommended for cancer survivors rather than patients undergoing treatment. It is essential to develop adapted, unsupervised, home-based PA programs to ensure access to PA for all cancer patients, particularly those living in rural areas or who have difficulty accessing healthcare. The PA program CREATE is a simple, unsupervised PA program based on patients' functional capacities. Depending on the patient's functional capacity, one of 7 PA programs will be prescribed by the doctor. The patient must perform the program independently for 6 months. Telephone follow-ups (weeks 1, 2, 4, 6, 9, 12, 16, 20, et 24) as well as a monthly in-person follow-up visit will be made to adjust the prescription.

ELIGIBILITY:
inclusion criteria:

* suffering from a hematological malignancy (Myelodysplasia, Leukemia of any type, Lymphoma, Myeloma)
* patient affiliated to a social security insurance
* Patient undergoing or scheduled chemotherapy (< 3 months) and/or immunotherapy and/or targeted therapy.

Exclusion criteria:

* Life expectancy estimated at less than 3 months by the unit doctor;
* Cognitive impairment (not allowing comprehension of the physical activity program and research project) defined by Mini-Mental State Examination (MMSE) <20/30;
* Patient included in a clinical trial that potentially interferes with the study objective (geriatric interventional study, early drug study, study modifying the patient's lifestyle habits).;
* Acute health problem (fever, severe anemia, intense pain, etc.) limiting the possibility of involvement in the program;
* Contraindication to physical activity;
* Patient under legal protection (guardianship or curatorship or safeguard of justice);
* Refusal of patient or primary caregiver to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: geriatric population suffering from a hematological malignancy (Myelodysplasia, Leukemia of any type, Lymphoma, Myeloma
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the PA program | 6 months
  PA program is considered feasible if at least 50% of them complete at least 70% of the prescribed sessions. Adherence is recorded in a logbook (every day), during the usual follow-up at the hospital (every month) and during telephone follow-up (weeks 1, 2, 4, 6, 9, 12, 16, 20, et 24).

CONTACTS AND LOCATIONS:
Overall Officials: Yves Rolland, Study Director — University Hospital, Toulouse
Locations (1):
- Chu de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided